CLINICAL TRIAL: NCT00179335
Title: Cross Sectional Case-Sectional Control Pharmacokinetic Study of Efavirenz or Lopinavir/Ritonavir as Part of an Antiretroviral Regimen With Two Nucleosides in HIV-Infected Adults 55 Years of Age or Older Compared With Adults Aged 18-35 Years
Brief Title: Comparative Pharmacokinetics (PK) Study of Efavirenz or Lopinavir/Ritonavir Between Older and Younger HIV-Infected Adults
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Abbott (Industry); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: CCI 03 143
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: HIV Infections
Keywords: Regular lopinavir/ritonavir or Efavirenz use; Age >/= 55 y or </= 35 y; HIV+
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Residual plasma left from measurement of drug levels.

INTERVENTIONS:
Procedure: Blood drawing to determine drug levels

SUMMARY:
HIV infected patients, aged </= 35 years and aged >/= 55 years, who are regularly taking either efavirenz (EFV) or lopinavir/ritonavir (Lop/r) as part of their antiretroviral regimen are being asked to spend 12 hours at the researchers' clinic (the ACS clinic at Jacobi Medical Center, Bronx, New York) for an intensive pharmacokinetic study in which 5 cc of blood will be drawn 9 times over a 12 hour period. Patients taking EFV will return for one additional blood draw the following day.

DETAILED DESCRIPTION:
HIV infected patients, aged </= 35 years and aged >/= 55 years, who are regularly taking either efavirenz or lopinavir/ritonavir as part of their antiretroviral regimen are being asked to spend 12 hours at our clinic (the ACS clinic at Jacobi Medical Center, Bronx, NY) for an intensive pharmacokinetic study in which 5 cc of blood will be drawn 9 times over a 12 hour period. Patients taking EFV will return for one additional blood draw the following day.

Patients will be asked to come to the clinic at 7 am and bring their medication to the clinic. Blood will be drawn to obtain a trough level of either EFV or Lop/r after which the patient will be instructed to take their EFV or Lop/r. Then blood will be drawn 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours later. Patients on EFV will be asked to return the next morning for a 24 hour blood level.

The blood will be spun and the plasma frozen at - 70 C. The plasma samples, labelled with the patients' initials and the draw date, will be shipped to University of Alabama, Department of Pharmacology, where the drug levels will be measured.

Patients will be recruited from the ACS outpatient clinic. They will be identified by their providers.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Taking lopinavir/ritonavir or efavirenz
* Age </= 35 years or >/= 55 years

Exclusion Criteria:

* Concurrent therapy with drugs that alter lopinavir/ritonavir levels.
* Other renal or kidney disease.
* Chronic hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pts enrolled in our clinic who are on either lopinavir/ritonavir or efavirenz, who are tolerating their HIV meds and who are judged to be compliant.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2003-08; Primary Completion 2006-01 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Jenny-Avital, MD, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine; Edward Acosta, Pharm D, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Jacobi Medical Center ACS Clinic, The Bronx, New York, United States